CLINICAL TRIAL: NCT01421316
Title: Reducing Hair Loss With Volumetric Arc Therapy in Patients Treated With Whole Brain Radiotherapy: a Phase II Trial
Brief Title: Hair-sparing Whole Brain Radiotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No reduction in hair loss 1 month after treatment
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011/504
Record Dates: First submitted 2011-08-17; First posted 2011-08-22 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Brain Metastases; Small Cell Lung Cancer
Keywords: Patients treated with whole brain radiotherapy in the setting of brain metastases; Patients treated with whole brain radiotherapy in the prophylactic treatment for small cell lung cancer (extended disease).
MeSH Terms: conditions — Brain Neoplasms; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Whole brain radiotherapy with volumetric arc therapy — Whole brain radiotherapy with volumetric arc therapy is used.

SUMMARY:
Up to 10% of patients with cancer will develop symptomatic brain metastases. Given this limited survival it is important to consider quality of life (QOL) when treating these patients. Whole brain radiotherapy (WBRT) can increase survival to 6 month. However, WBRT itself has been shown to reduce QOL by increasing drowsiness, leg weakness and hair loss in patients with brain metastases. Both fatigue and hair loss were reported to have the largest decline in QOL scores when WBRT is used in the prophylactic setting in small cell lung cancer. Recent technological improvements in patient positioning and treatment planning will allow us to treat the whole brain with reduced margins, allowing better sparing of the scalp. In view of the large impact of hair loss on quality of life, the investigators hypothesize to see an improved quality of life with scalp sparing techniques.

Study hypothesis: Volumetric arc therapy results in a reduced hair loss and a subsequent clinically important improvement in QOL.

ELIGIBILITY:
Inclusion Criteria:

* Brain metastases
* Age ≥ 18 years.
* Signed informed consent
* Recursive Partitioning Analysis (RPA) class III patients
* Recursive Partitioning Analysis (RPA) class I-II patients and >3 brain metastases
* Patients with small cell lung cancer extended disease eligible for prophylactic Whole-Brain Radiotherapy (WBRT).

Exclusion Criteria:

* Previous whole brain radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The European Organization for Research and Treatment of Cancer (EORTC)quality of life questionnaire (C15-PAL and BN20) measured at 1 month following treatment. | At 1 month.
  Quality of life questionnaires are used.

SECONDARY OUTCOMES:
Hair quality before treatment and at 1 month following treatment. | at 1 month following treatment
  Key measurements: trichogram are used.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Belgium, Ghent, Belgium